CLINICAL TRIAL: NCT05749939
Title: Brief Online Acceptance Commitment Therapy for Caregivers: a Fully Longitudinal Mixed Methods RC
Brief Title: Acceptance Commitment Therapy for Caregivers of People with Memory Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Audrey Juhasz, Principal Investigator, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13040
Record Dates: First submitted 2023-01-26; First posted 2023-03-01 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Caregiver Burden; Behavioral and Psychiatric Symptoms of Dementia; Depressive Symptoms; Quality of Life; Psychological Flexibility; Sleep Quality; Positive Aspects of Caregiving
Keywords: Acceptance and Commitment Therapy; Caregivers of people with dementia
MeSH Terms: conditions — Caregiver Burden; Behavior; Depression; Sleep Initiation and Maintenance Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Randomized wait list control trial. Participants are assigned to treatment and wait list groups. Wait list participants receive treatment after 4 weeks of waiting. Treatment participants receive treatment immediately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Receives access to the online ACT course immediately after enrollment
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Waitlist (No Intervention): Receives access to the online ACT course 30 days after enrollment

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and commitment therapy (ACT) combines the skills of acceptance, cognitive defusion, being present, self as context, values, and committed action to help individuals engage with a meaningful life. A goal of ACT is to help people develop psychological flexibility, meaning they can experience and live with difficult thoughts and emotions, and still pursue what matters to them. The current project is an online, self-guided, 6-session intervention. Each session is expected to take about 30 minutes each, and the entire course will take approximately 3-4 weeks to complete, as users are encouraged to take a few days in between sessions. Within each session, participants will read about concepts and ACT metaphors, apply ACT concepts to general and care- specific vignettes, and apply ACT concepts to their own lives and care situations. Interactive experiences are included in each session and ends with a printable summary with practice skills before proceeding.
  Arms: Treatment

SUMMARY:
Family caregivers for persons with dementia report high levels of depression, stress, and burden. Caregivers' limited time, transportation constraints, and unpredictable schedules make on-line, self-guided interventions more accessible and scalable. Acceptance and Commitment Therapy (ACT) is an established and effective in-person therapy, well-suited to the dementia care giving context where caregivers cannot minimize stress exposure, and report difficult thoughts and emotions. ACT for Caregivers is an on-line self-guided ACT intervention that showed effectiveness in a Stage I pilot (n=52) with participants reporting decreased depressive symptoms, stressful reactions to caring, and caregiver burden, and increased quality of life and positive aspects of caring (all p <.05). Learning from the pilot, the current Stage III intervention will shorten the program from 10 sessions to 6 sessions. The investigators introduce a wait list randomized control trial (RCT) design with fully longitudinal mixed methods to evaluate ACT for Caregivers. Data will be collected at pretest, post-test, and 6-weeks follow-up. Study aims are: 1) to evaluate ACT for Caregivers in a larger sample using an RCT, 2) to understand user experiences and the process of change by collecting short response data from all participants at all time points and interviewing a subset of participants in-depth at two time points, 3) to integrate quantitative and qualitative findings and examine areas of convergence and divergence. This project offers a promising prevention and intervention program to support family caregivers that is scalable, at low cost and with high impact.

DETAILED DESCRIPTION:
Literature Review An estimated 6.2 million Americans live with Alzheimer's disease or a related dementia (ADRD), and over 11 million family caregivers currently assist a person with ADRD. The combination of cognitive impairment, behavioral symptoms, and loss of a reciprocal relationship can be very challenging for caregivers. Chronic stress can affect caregivers' mental and physical health, and sometimes lead to lower quality of care for the person with ADRD. Research indicates promising pathways to support caregiver mental health through interventions that address coping skills, self-care, and commitment to personal values.

A growing number of studies demonstrate that Acceptance and Commitment Therapy (ACT) is effective in reducing distress across a broad number of conditions and contexts. ACT combines the skills of acceptance, cognitive defusion, being present, self as context, values, and committed action to help individuals engage with a meaningful life. ACT helps individuals feel less guided by rigid or critical thoughts, and it teaches individuals to be nonjudgmental and present when difficult experiences arise. A goal of ACT is to help people develop psychological flexibility, meaning being capable of experiencing and living with difficult thoughts and emotions, while still pursue what matters to the individual.

Caregivers of persons with ADRD often disconnect from meaningful activities and relationships due to the ongoing supervision needed for their loved one. Caregivers experience feelings of grief and loss, even while their loved one is still alive, and sometimes use avoidant approaches to minimize feelings of loss, guilt, and exhaustion. ACT with a therapist is highly effective in helping family caregivers of persons with ADRD to reduce depression, anxiety, and experiential avoidance.

While ACT is traditionally delivered in person with a trained therapist, it has also demonstrated effective psychological and emotional benefits in an online format. Online interventions are well-suited for dementia caregivers, who have limited time, transportation constraints, and unpredictable care schedules. Online programs can be accessed conveniently around care routines, do not require driving or finding supervision for the care receiver, are low-cost for users and providers, and are able to relay informational, emotional, and task-specific support, even to hard-to-reach populations, such as those living in rural areas. Clinical trials indicate that online therapy is effective, arguably equally effective to face-to-face therapy.

The Current Study In 2021, USU researchers published results of a pilot study for an online, self-guided ACT for Caregivers of persons with ADRD. Participation in this 10-session online intervention was associated with decreased depressive symptoms, care-related burden, and stress reactions to behavioral symptoms. Caregivers also reported increased positive aspects of caregiving and quality of life. Importantly, the pilot study lacked a control condition. There is also increasing evidence that ACT, can be delivered more concisely; ACT research in other populations suggests a brief approach may be equally effective as longer programs. Given the time constraints of this population, shorter programs may be more appealing for users. The primary aim of the current project is to use a randomized waitlist controlled trial design to determine whether a shorter six session ACT intervention is effective in improving relevant caregiver outcomes.

While the 2021 pilot demonstrated that ACT could improve caregivers outcomes, the investigators were unable to examine the specific ways that participants utilized ACT in their lives. In other words, currently the field recognizes that individuals can change, but knows less about the mechanisms of change, which is important in moving these interventions forward, and on a larger scale. A mixed methods design will allow for the examination of this project's second aim to integrate participants' quantitative data with descriptions of their lived experience to better understand how the intervention promotes positive change.

Research Objectives The current study uses a randomized wait-list controlled trial design and fully longitudinal mixed methods analysis to examine the effectiveness of a condensed online ACT for Caregivers program.

Aim 1: Empirically evaluate the effectiveness of a six-session online ACT intervention in reducing negative aspects of caregiving (depressive symptoms, burden, stressful reactions to memory and behavior problems) and promotion of positive thoughts and behaviors (recognition of positive aspects of caregiving, improved sleep quality, and increased quality of life).

Aim 2: Qualitatively explore caregivers' lived experience with the intervention and ways that caregivers are applying the skills in their lives and examine the extent to which caregivers' descriptions align with and expand on theory-based mechanisms of change.

Impact

Anticipated Outcomes

The anticipated outcomes of our study are:

1. to improve wellbeing of 100 family caregivers for persons with ADRD via an online, self- guided intervention
2. to complete a Stage III study with sufficient methodological rigor to provide evidence of program effectiveness and justify more widespread implementation of this program.
3. to produce necessary documentation of effectiveness to support pursuit of further funding through the National Institute of Health (NIH) or the National Institute of Mental Health (NIMH). NIH expects to spend 3.4+ billion in ADRD grants in the next year.
4. to understand how caregivers' experience changes over time within and following an intervention
5. to understand how ACT-based skills act as potential drivers of change for family caregivers.

Implications Our study is a robust Stage III test of the effectiveness of a shorter (more user-friendly) version of ACT for Caregivers, which has not yet been empirically tested using a randomized control design. While evidence suggests that ACT in other populations can be delivered effectively in as little as one face-to- face session, little is known about the 'dosage' required for online, self-guided interventions. If our shorter ACT for Caregivers protocol is effective in improving caregiver outcomes, the program will move forward towards the implementation goal of being offered for free (or at very low cost) through Utah State University's Alzheimer's Research Center.

The ACT for Caregivers Stage I pilot study (with the longer 10-session format) demonstrated improved outcomes but inadequate power to examine more nuanced mechanisms for change, and without qualitative data collected. With a larger sample, the present study allows for adequate power to examine change mechanisms quantitatively. Qualitative interviews and mixed methods approaches are added to the current study to understand change, and how ACT-related skills contribute to change. Although fully longitudinal mixed methods research is becoming more common in health research, it is still novel in program development and evaluation with ADRD caregivers. Fully longitudinal mixed methods research allows for a holistic examination of whether and how change occurs over time and is therefore highly relevant for evaluating promising intervention programs in the growing population of family caregivers for persons with ADRD.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identification as a family caregiver to a person with dementia or other significant memory loss
2. Interest in taking part in an on-line self-guided program with multiple assessments up through 6-week follow-up
3. Distressed from the care giving role, as measured by a score of 4+ on a single item "How distressed are you by caring for your family member?" (1 not at all to 10 extremely)
4. Ability to read/write English
5. Access to a computer/smartphone/tablet with Internet
6. Caregiver does not have to live with the care recipient, as distress can arise with or without cohabitation, participants must live within the United States.

Exclusion Criteria:

1. Not caring for a family caregiver to a person with dementia or other significant memory loss
2. Not interested in an on-line self-guided program with multiple assessments up through 6-week follow-up
3. Responds with a score of 3 or less when asked "How distressed are you by caring for your family member?" (1 not at all to 10 extremely)
4. Inability to read/write English
5. Does not have reliable access to a computer/smartphone/tablet with Internet.
6. Lives outside of the United States
7. Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Mean group (waitlist/treatment) differences in caregiver burden | 30 days
  Group differences between waitlist and treatment group scores after the treatment group has had access to the treatment for 30 days and the waitlist group has not received any intervention for the same amount of time. Caregiver burden is measured by a 12-item [short] caregiver burden scale. Participants rate the impact of caregiving on multiple aspects of health (response range 0 never to 4 nearly always). A total possible summed scores range from 0 to 48; higher scores indicate higher burden.
Mean group (waitlist/treatment) differences in depressive symptoms | 30 days
  Group differences between waitlist and treatment group scores after the treatment group has had access to the treatment for 30 days and the waitlist group has not received any intervention for the same amount of time. Depressive symptoms are measured by 10-item [short] Center for Epidemiological Studies Depression Scale (CES-D). Participants rate the frequency of depressive symptoms during the past week. Responses range from 1 rarely or none of the time to 4 all of the time, with possible summed scores ranging from 10 to 40; higher scores indicate more depressive symptoms.
Mean group (waitlist/treatment) differences in positive aspects of caregiving | 30 days
  Group differences between waitlist and treatment group scores after the treatment group has had access to the treatment for 30 days and the waitlist group has not received any intervention for the same amount of time. Positive aspects of caregiving will be measured using a 9-item Positive Aspects of Caregiving measure. Items use the following stem "Providing help to (name) has…", with example items such as "made me feel useful" and "enabled me to appreciate life more." Responses range from 1 disagree a lot to 5 agree a lot, and items are summed with a possible score range from 9 to 45; higher scores indicate more positive aspects of caregiving.
Mean group (waitlist/treatment) differences in sleep quality | 30 days
  Group differences between waitlist and treatment group scores after the treatment group has had access to the treatment for 30 days and the waitlist group has not received any intervention for the same amount of time. Sleep quality will be measured by a 1-item Sleep Quality Scale ranging from 0 terrible to 10 excellent, with higher scores indicating higher quality. Respondents are asked to consider the overall quality of sleep on most nights over the last seven days only.
Mean group (waitlist/treatment) differences in psychological flexibility | 30 days
  Group differences between waitlist and treatment group scores after the treatment group has had access to the treatment for 30 days and the waitlist group has not received any intervention for the same amount of time. Psychological flexibility will be measured by the 23-item CompACT consisting of three subscales: openness to experience (10 items; possible score range 0 to 60), behavioral awareness (5 items; possible score range 0 to 30), and valued actions (8 items; possible score range 0 to 48). Responses range from 0 strongly disagree to 6 strongly agree. Some items are reverse scored. Lower scores indicate more psychological flexibility.
Mean group (waitlist/treatment) differences in quality of life | 30 days
  Group differences between waitlist and treatment group scores after the treatment group has had access to the treatment for 30 days and the waitlist group has not received any intervention for the same amount of time. Quality of life will be measured by a 1-item visual analogue scale ranging from 0 to 100, with higher scores indicating higher quality of life.
Within person change from Pretest measures at Posttest and Follow up in caregiver burden | Pretest before intervention, 30 days of treatment access, and 6 weeks after initial 30 day period
  Change over time for all participants comparing scores from before the intervention, to after 30 day of access to the treatment, and again 6 weeks after the end of the initial 30 day period. Caregiver burden is measured by a 12-item [short] caregiver burden scale. Participants rate the impact of caregiving on multiple aspects of health (response range 0 never to 4 nearly always). A total possible summed scores range from 0 to 48; higher scores indicate higher burden.
Within person change from Pretest measures at Posttest and Follow up in depressive symptoms | Pretest before intervention, 30 days of program access, and 6 weeks after initial 30 day period
  Change over time for all participants comparing changes in scores from before the intervention, to after 30 day of access to the treatment, and again 6 weeks after the end of the initial 30 day period. Depressive symptoms are measured by 10-item [short] Center for Epidemiological Studies Depression Scale (CES-D). Participants rate the frequency of depressive symptoms during the past week. Responses range from 1 rarely or none of the time to 4 all of the time, with possible summed scores ranging from 10 to 40; higher scores indicate more depressive symptoms.
Within person change from Pretest measures at Posttest and Follow up in positive aspects of caregiving | Pretest before intervention, 30 days of program access, and 6 weeks after initial 30 day period
  Change over time for all participants comparing changes in scores from before the intervention, to after 30 day of access to the treatment, and again 6 weeks after the end of the initial 30 day period. Positive aspects of caregiving will be measured using a 9-item Positive Aspects of Caregiving measure. Items use the following stem "Providing help to (name) has…", with example items such as "made me feel useful" and "enabled me to appreciate life more." Responses range from 1 disagree a lot to 5 agree a lot, and items are summed with a possible score range from 9 to 45; higher scores indicate more positive aspects of caregiving.
Within person change from Pretest measures at Posttest and Follow up in sleep quality | Pretest before intervention, 30 days of program access, and 6 weeks after initial 30 day period
  Change over time for all participants comparing changes in scores from before the intervention, to after 30 day of access to the treatment, and again 6 weeks after the end of the initial 30 day period. Sleep quality will be measured by a 1-item Sleep Quality Scale ranging from 0 terrible to 10 excellent, with higher scores indicating higher quality. Respondents are asked to consider the overall quality of sleep on most nights over the last seven days only.
Within person change from Pretest measures at Posttest and Follow up in psychological flexibility | Pretest before intervention, 30 days of program access, and 6 weeks after initial 30 day period
  Change over time for all participants comparing changes in scores from before the intervention, to after 30 day of access to the treatment, and again 6 weeks after the end of the initial 30 day period. Psychological flexibility will be measured by the 23-item CompACT consisting of three subscales: openness to experience (10 items; possible score range 0 to 60), behavioral awareness (5 items; possible score range 0 to 30), and valued actions (8 items; possible score range 0 to 48). Responses range from 0 strongly disagree to 6 strongly agree. Some items are reverse scored. Lower scores indicate more psychological flexibility.
Within person change from Pretest measures at Posttest and Follow up in quality of life | Pretest before intervention, 30 days of program access, and 6 weeks after initial 30 day period
  Change over time for all participants comparing changes in scores from before the intervention, to after 30 day of access to the treatment, and again 6 weeks after the end of the initial 30 day period. Quality of life will be measured by a 1-item visual analogue scale ranging from 0 to 100, with higher scores indicating higher quality of life.
Description of participant experience using this intervention | 30 days
  Qualitative interviews will capture how participant experiences support, refine, and contradict acceptance commitment therapy (ACT) principles.
Change from Post intervention experience at Follow up | 30 days after access to program to 6 weeks later
  Qualitative interviews will capture changes in participant's attitudes and enactment of principles learned during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey C Juhasz, PhD, Principal Investigator — Utah State University; Elizabeth Fauth, PhD, Study Director — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Dr. Elizabeth Fauth will review requests and criteria.

REFERENCES:
- [Background] Fauth EB, Novak JR, Levin ME. Outcomes from a pilot online Acceptance and Commitment Therapy program for dementia family caregivers. Aging Ment Health. 2022 Aug;26(8):1620-1629. doi: 10.1080/13607863.2021.1942432. Epub 2021 Jul 7. PMID 34233133
- [Background] Plano Clark VL, Anderson N, Wertz JA, Zhou Y, Schumacher K, & Miaskowski C. Conceptualizing longitudinal mixed methods designs: A methodological review of health sciences research. Journal of Mixed Methods Research. 2015; 9(4): 297-319.
- [Background] Dochat C, Wooldridge JS, Herbert MS, Lee MW, Afari N. Single-Session Acceptance and Commitment Therapy (ACT) Interventions for Patients with Chronic Health Conditions: A Systematic Review and Meta-Analysis. J Contextual Behav Sci. 2021 Apr;20:52-69. doi: 10.1016/j.jcbs.2021.03.003. Epub 2021 Mar 6. PMID 33868913
- [Background] Cuijpers P, Donker T, van Straten A, Li J, Andersson G. Is guided self-help as effective as face-to-face psychotherapy for depression and anxiety disorders? A systematic review and meta-analysis of comparative outcome studies. Psychol Med. 2010 Dec;40(12):1943-57. doi: 10.1017/S0033291710000772. Epub 2010 Apr 21. PMID 20406528
- [Background] Godwin KM, Mills WL, Anderson JA, Kunik ME. Technology-driven interventions for caregivers of persons with dementia: a systematic review. Am J Alzheimers Dis Other Demen. 2013 May;28(3):216-22. doi: 10.1177/1533317513481091. Epub 2013 Mar 25. PMID 23528881
- [Background] Bayly M, Morgan D, Froehlich Chow A, Kosteniuk J, Elliot V. Dementia-Related Education and Support Service Availability, Accessibility, and Use in Rural Areas: Barriers and Solutions. Can J Aging. 2020 Dec;39(4):545-585. doi: 10.1017/S0714980819000564. Epub 2020 Jan 24. PMID 31975685
- [Background] Ng GT. Support for family caregivers: what do service providers say about accessibility, availability and affordability of services? Health Soc Care Community. 2009 Nov;17(6):590-8. doi: 10.1111/j.1365-2524.2009.00858.x. Epub 2009 May 13. PMID 19469918
- [Background] Brown M, Glendenning A, Hoon AE, John A. Effectiveness of Web-Delivered Acceptance and Commitment Therapy in Relation to Mental Health and Well-Being: A Systematic Review and Meta-Analysis. J Med Internet Res. 2016 Aug 24;18(8):e221. doi: 10.2196/jmir.6200. PMID 27558740
- [Background] Levin ME, Pistorello J, Seeley JR, Hayes SC. Feasibility of a prototype web-based acceptance and commitment therapy prevention program for college students. J Am Coll Health. 2014;62(1):20-30. doi: 10.1080/07448481.2013.843533. PMID 24313693
- [Background] Coon DW, Thompson L, Steffen A, Sorocco K, Gallagher-Thompson D. Anger and depression management: psychoeducational skill training interventions for women caregivers of a relative with dementia. Gerontologist. 2003 Oct;43(5):678-89. doi: 10.1093/geront/43.5.678. PMID 14570964
- [Background] Han A, Yuen HK, Jenkins J. Acceptance and commitment therapy for family caregivers: A systematic review and meta-analysis. J Health Psychol. 2021 Jan;26(1):82-102. doi: 10.1177/1359105320941217. Epub 2020 Jul 10. PMID 32659142
- [Background] Losada A, Marquez-Gonzalez M, Romero-Moreno R. Mechanisms of action of a psychological intervention for dementia caregivers: effects of behavioral activation and modification of dysfunctional thoughts. Int J Geriatr Psychiatry. 2011 Nov;26(11):1119-27. doi: 10.1002/gps.2648. Epub 2010 Nov 9. PMID 21061414
- [Background] Losada A, Marquez-Gonzalez M, Romero-Moreno R, Mausbach BT, Lopez J, Fernandez-Fernandez V, Nogales-Gonzalez C. Cognitive-behavioral therapy (CBT) versus acceptance and commitment therapy (ACT) for dementia family caregivers with significant depressive symptoms: Results of a randomized clinical trial. J Consult Clin Psychol. 2015 Aug;83(4):760-72. doi: 10.1037/ccp0000028. Epub 2015 Jun 15. PMID 26075381
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Coen RF, O'Boyle CA, Coakley D, Lawlor BA. Individual quality of life factors distinguishing low-burden and high-burden caregivers of dementia patients. Dement Geriatr Cogn Disord. 2002;13(3):164-70. doi: 10.1159/000048648. PMID 11893838
- [Background] Gao C, Chapagain NY, Scullin MK. Sleep Duration and Sleep Quality in Caregivers of Patients With Dementia: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Aug 2;2(8):e199891. doi: 10.1001/jamanetworkopen.2019.9891. PMID 31441938
- [Background] Li R, Cooper C, Livingston G. Relationship of coping style to mood and anxiety disorders in dementia carers. Curr Opin Psychiatry. 2014 Jan;27(1):52-6. doi: 10.1097/YCO.0000000000000020. PMID 24270483
- [Background] Romero-Moreno R, Losada A, Marquez-Gonzalez M, Mausbach BT. Stressors and anxiety in dementia caregiving: multiple mediation analysis of rumination, experiential avoidance, and leisure. Int Psychogeriatr. 2016 Nov;28(11):1835-1844. doi: 10.1017/S1041610216001009. Epub 2016 Jul 26. PMID 27457894
- [Background] Walter E, Pinquart M. How Effective Are Dementia Caregiver Interventions? An Updated Comprehensive Meta-Analysis. Gerontologist. 2020 Nov 23;60(8):609-619. doi: 10.1093/geront/gnz118. PMID 33226434
- [Background] Chiao CY, Wu HS, Hsiao CY. Caregiver burden for informal caregivers of patients with dementia: A systematic review. Int Nurs Rev. 2015 Sep;62(3):340-50. doi: 10.1111/inr.12194. Epub 2015 Jun 8. PMID 26058542
- [Background] Finkel S. Introduction to behavioural and psychological symptoms of dementia (BPSD). Int J Geriatr Psychiatry. 2000 Jul;15 Suppl 1:S2-4. doi: 10.1002/(sici)1099-1166(200004)15:1+3.0.co;2-3. No abstract available. PMID 10767742
- [Background] Alzheimer's Association (2021). Alzheimer's disease facts and figures 2021. Retrieved from https://www.alz.org/alzheimers-dementia/facts-figures Oct 5, 2022.
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Tarlow BJ, Wisniewski SR, Belle SH, Rubert M, Ory MG, & Gallagher-Thompson D. Positive Aspects of Caregiving: Contributions of the REACH Project to the Development of New Measures for Alzheimer's Caregiving. Research on Aging. 2004; 26(4): 429-453. doi:10.1177/0164027504264493
- [Background] Snyder E, Cai B, DeMuro C, Morrison MF, Ball W. A New Single-Item Sleep Quality Scale: Results of Psychometric Evaluation in Patients With Chronic Primary Insomnia and Depression. J Clin Sleep Med. 2018 Nov 15;14(11):1849-1857. doi: 10.5664/jcsm.7478. PMID 30373688
- [Background] Lowenberg B, van Putten WL, Ferrant A, Ossenkoppele G, Vellenga E, Verdonck LF, Gratwohl A, Boogaerts MA. Peripheral blood progenitor cell transplantation as an alternative to autologous marrow transplantation in the treatment of acute myeloid leukemia. Stem Cells. 1997;15 Suppl 1:177-80; discussion 181. doi: 10.1002/stem.5530150823. PMID 9368339
- [Background] de Boer AG, van Lanschot JJ, Stalmeier PF, van Sandick JW, Hulscher JB, de Haes JC, Sprangers MA. Is a single-item visual analogue scale as valid, reliable and responsive as multi-item scales in measuring quality of life? Qual Life Res. 2004 Mar;13(2):311-20. doi: 10.1023/B:QURE.0000018499.64574.1f. PMID 15085903